CLINICAL TRIAL: NCT04580602
Title: Correlation Between Bleeding Complication and Treatment Failure on P2Y12 Inhibitors and Its Predictions Based on Cipherome's Pharmacogenomic Technology
Brief Title: Association Between Genetic Variant Scores and P2Y12 Inhibitor Effects
Acronym: CARES1
Status: Completed | Type: Observational
Sponsor: Cipherome, Inc. (Industry)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: C03-001 BD002
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Stent Thrombosis; Ischemic Stroke; Myocardial Infarction; Acute Coronary Syndrome
MeSH Terms: conditions — Ischemic Stroke; Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Laboratory blood draw
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ADR Group: Major Bleeding BARC Bleeding Criteria Type 2,3,5
- Control Group: No ADR or treatment failure, case-control matched to experimental groups
- Treatment Failure Group: Major Adverse Cardiovascular Events (MACE)

SUMMARY:
The goal of this study is to predict and prevent adverse drug events by investigating the impact of genetic variants, demographics, and environmental factors in subjects status post myocardial infarction and percutaneous coronary insertion who have experienced adverse drug events while on P2Y12 inhibitors.

DETAILED DESCRIPTION:
The goal of this study it to validate Cipherome's drug safety score (DSS) in its predictive accuracy for severe adverse drug reactions (ADRs). The DSS is calculated on a scale of 0 to 1, with preliminary studies demonstrating that scores below 0.3 correlated with a higher chance of an ADR and scores above 0.7 correlated with a lower chance of an ADR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years and older, who are on P2Y12 inhibitors (clopidogrel, prasugrel, or ticagrelor).
2. Ability to provide informed consent.

Exclusion Criteria:

1. Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects (status post myocardial infarction and percutaneous coronary insertion) who have experienced adverse drug events while on P2Y12 inhibitors in order to improve future prediction and prevention of adverse events.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
To assess the predictive accuracy of Cipherome's drug safety score (DSS) in correlating with serious ADRs in subjects on P2Y12 inhibitors. | Within 24 months of clopidogrel therapy initiation
  The primary endpoint is to assess the predictive accuracy of the DSS compared to actual clinical outcomes of treatment failure (major adverse cardiovascular events or MACE) or bleeding (per BARC criteria) in subjects on P2Y12 inhibitors. The DSS is calculated on a scale of 0 to 1, with preliminary studies demonstrating that scores below 0.3 correlated with a higher chance of an ADR and scores above 0.7 correlated with a lower chance of an ADR.

SECONDARY OUTCOMES:
To assess the predictive accuracy of the DSS in correlating with serious ADRs compared to clinical guidelines (e.g., Clinical Pharmacogenetics Implementation Consortium (CPIC)) in subjects on P2Y12 inhibitors. | Within 24 months of clopidogrel therapy initiation
  The secondary endpoint is to assess the predictive accuracy of the DSS compared to current evidence-based clinical guidelines, such as CPIC, for serious ADRs (e.g., treatment failure such as MACE) for subjects on P2Y12 inhibitors.
To assess the predictive accuracy of the DSS in correlating with major bleeding compared to clinical guidelines (CPIC) in subjects on P2Y12 inhibitors. | Within 24 months of clopidogrel therapy initiation
  The secondary endpoint is to assess the predictive accuracy of the DSS compared to CPIC, for major bleeding per BARC criteria, in subjects on P2Y12 inhibitors.

OTHER OUTCOMES:
To discover novel pharmacogenetic variants associated with P2Y12 metabolism. | Within 24 months of clopidogrel therapy initiation
  We will assess the DSS within genes and evaluate the genetic-pathways for P2Y12 metabolism. Novel variants will be assessed using whole genome sequencing to evaluate the genetic pathways in individuals with serious ADRs and treatment failures. Through our analyses we intend to identify novel genetic variants in subjects with serious ADRs or treatment failure while on P2Y12 inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: Jungwon Suh, MD, Principal Investigator — SNUBH
Locations (1):
- SNUBH, Seongnam-si, Gyonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pereira NL, Rihal CS, So DYF, Rosenberg Y, Lennon RJ, Mathew V, Goodman SG, Weinshilboum RM, Wang L, Baudhuin LM, Lerman A, Hasan A, Iturriaga E, Fu YP, Geller N, Bailey K, Farkouh ME. Clopidogrel Pharmacogenetics. Circ Cardiovasc Interv. 2019 Apr;12(4):e007811. doi: 10.1161/CIRCINTERVENTIONS.119.007811. PMID 30998396
- [Background] Pan Y, Chen W, Xu Y, Yi X, Han Y, Yang Q, Li X, Huang L, Johnston SC, Zhao X, Liu L, Zhang Q, Wang G, Wang Y, Wang Y. Genetic Polymorphisms and Clopidogrel Efficacy for Acute Ischemic Stroke or Transient Ischemic Attack: A Systematic Review and Meta-Analysis. Circulation. 2017 Jan 3;135(1):21-33. doi: 10.1161/CIRCULATIONAHA.116.024913. Epub 2016 Nov 2. PMID 27806998
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083
- [Background] Jeong YH, Tantry US, Kim IS, Koh JS, Kwon TJ, Park Y, Hwang SJ, Bliden KP, Kwak CH, Hwang JY, Gurbel PA. Effect of CYP2C19*2 and *3 loss-of-function alleles on platelet reactivity and adverse clinical events in East Asian acute myocardial infarction survivors treated with clopidogrel and aspirin. Circ Cardiovasc Interv. 2011 Dec 1;4(6):585-94. doi: 10.1161/CIRCINTERVENTIONS.111.962555. Epub 2011 Nov 1. PMID 22045970
- [Background] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Background] Park KH, Jeong MH, Kim HK, Ahn TH, Seung KB, Oh DJ, Choi DJ, Kim HS, Gwon HC, Seong IW, Hwang KK, Chae SC, Kim KB, Kim YJ, Cha KS, Oh SK, Chae JK; KAMIR-NIH Registry Investigators. Comparison of prasugrel versus clopidogrel in Korean patients with acute myocardial infarction undergoing successful revascularization. J Cardiol. 2018 Jan;71(1):36-43. doi: 10.1016/j.jjcc.2017.05.003. Epub 2017 Jun 30. PMID 28673508
- [Background] Park DW, Kwon O, Jang JS, Yun SC, Park H, Kang DY, Ahn JM, Lee PH, Lee SW, Park SW, Choi SW, Lee SG, Yoon HJ, Ahn T, Kim MH, Nah DY, Lee SY, Chae JK, Park SJ; TICAKOREA Investigators. Clinically Significant Bleeding With Ticagrelor Versus Clopidogrel in Korean Patients With Acute Coronary Syndromes Intended for Invasive Management: A Randomized Clinical Trial. Circulation. 2019 Dec 3;140(23):1865-1877. doi: 10.1161/CIRCULATIONAHA.119.041766. Epub 2019 Sep 25. PMID 31553203
- [Background] Parks AL, Fang MC. Scoring Systems for Estimating the Risk of Anticoagulant-Associated Bleeding. Semin Thromb Hemost. 2017 Jul;43(5):514-524. doi: 10.1055/s-0037-1598061. Epub 2017 Mar 30. PMID 28359135
- [Background] Kang J, Park KW, Ki YJ, Park J, Rhee T, Kim CH, Han JK, Yang HM, Kang HJ, Koo BK, Nakamura M, Hamasaki T, Yokoi H, Cohen D, Kim HS. Development and Validation of an Ischemic and Bleeding Risk Evaluation Tool in East Asian Patients Receiving Percutaneous Coronary Intervention. Thromb Haemost. 2019 Jul;119(7):1182-1193. doi: 10.1055/s-0039-1688792. Epub 2019 May 12. PMID 31079414
- [Background] Claassens DMF, Vos GJA, Bergmeijer TO, Hermanides RS, van 't Hof AWJ, van der Harst P, Barbato E, Morisco C, Tjon Joe Gin RM, Asselbergs FW, Mosterd A, Herrman JR, Dewilde WJM, Janssen PWA, Kelder JC, Postma MJ, de Boer A, Boersma C, Deneer VHM, Ten Berg JM. A Genotype-Guided Strategy for Oral P2Y12 Inhibitors in Primary PCI. N Engl J Med. 2019 Oct 24;381(17):1621-1631. doi: 10.1056/NEJMoa1907096. Epub 2019 Sep 3. PMID 31479209
- [Background] Urban P, Mehran R, Colleran R, Angiolillo DJ, Byrne RA, Capodanno D, Cuisset T, Cutlip D, Eerdmans P, Eikelboom J, Farb A, Gibson CM, Gregson J, Haude M, James SK, Kim HS, Kimura T, Konishi A, Laschinger J, Leon MB, Magee PFA, Mitsutake Y, Mylotte D, Pocock S, Price MJ, Rao SV, Spitzer E, Stockbridge N, Valgimigli M, Varenne O, Windhoevel U, Yeh RW, Krucoff MW, Morice MC. Defining high bleeding risk in patients undergoing percutaneous coronary intervention: a consensus document from the Academic Research Consortium for High Bleeding Risk. Eur Heart J. 2019 Aug 14;40(31):2632-2653. doi: 10.1093/eurheartj/ehz372. PMID 31116395
- See also: Plavix package insert. (accessed March 26, 2020) — https://www.accessdata.fda.gov/drugsatfda_docs/label/2010/020839s048lbl.pdf